CLINICAL TRIAL: NCT06236113
Title: Low Dose Ketamine for Blunt Thoracic Trauma: A Prospective Randomized Trial
Brief Title: Low Dose Ketamine for Blunt Thoracic Trauma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Memorial Health Care (Other)
Responsible Party: Principal Investigator, Michaela A West, Trauma Research Chair, North Memorial Health Care
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04/18/46
Record Dates: First submitted 2024-01-12; First posted 2024-02-01 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Blunt Injury of Thorax; Multiple Rib Fractures, Involving Three Ribs
Keywords: Blunt Thoracic Trauma
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blinded, placebo-controlled study comparing saline infusion with low-dose ketamine versus saline infusion alone.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacist prepares medications for patients. Medication or placebo appear identical and are released to bedside nurse with weight based infusion instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo/Control (Placebo Comparator): Pharmacist will check randomization schedule. For placebo/control subject they will prepare an infusion bag of saline with no added medication. The Study Drug Bag will be released with a label that includes: Name of Study, Study Subject #, Patient (Pt) Name, Pt Medical record number (MR#), Pt Date of birth (DOB), and INFUSION RATE.
  Interventions: Drug: Ketamine 1 Mg/mL-NaCl 0.9% Intravenous Solution
- Low Dose Ketamine Infusion (LDKI) (Experimental): Infusion Bag will receive 100 mg of ketamine (Ketamine Infusion Subject). The Study Drug Bag will be released with a label that includes: Name of Study, Study Subject #, Patient Name, Pt MR#, Pt DOB, and INFUSION RATE. (Note: infusion rate is 0.1 mg/kg/hr and concentration of standard ketamine infusion bag is 1 mg/mL. That is, 100 mg of ketamine added to 100 mL saline).
  Interventions: Drug: Ketamine 1 Mg/mL-NaCl 0.9% Intravenous Solution

INTERVENTIONS:
Drug: Ketamine 1 Mg/mL-NaCl 0.9% Intravenous Solution — administered at rate of 0.1 mg/kg/hr
  Other Names: Low Dose Ketamine Infusion; Ketamine Drip

SUMMARY:
The goal of this Randomized controlled double-blinded trial is to compare the addition of a ketamine infusion to placebo, when added to standard care in adult blunt trauma patients with multiple rib fractures. The main question it aims to answer are: • addition of low dose ketamine infusion (LDKI) decreases narcotic use • does LDKI impact pulmonary complications, readmission, or hospital length of stay Participants will receive usual standard of care with up to 48 hours of LDKI or placebo. If there is a comparison group: Researchers will compare infusion of a saline infusion to LDKI to see if LDKI decreases need for narcotic analgesics use.

DETAILED DESCRIPTION:
Study Design: Randomized controlled double-blinded trial: Patients will then be randomized into one of two study groups. Both groups will receive a normal saline infusion for 48 hours of therapy. The treatment group will have ketamine added to their saline infusion via blinded pharmacy protocol to receive continuous infusion of ketamine at 0.1mg/kg/hour. The control group will receive only normal saline. Administration will occur via piggyback infusion in accordance with nursing policy.

Setting/Participants:

* North Memorial Health Hospital: patients on 5-South - Trauma Neuro Intensive Care Unit (TNICU) and 6-West - Trauma Floor
* 50 people will take part in this study. 25 study subjects will receive an infusion of ketamine and 25 will receive a saline infusion.
* Patients 18 years of age or older with 3 or more rib fractures admitted to North Memorial Health Hospital will be considered for the study.

Study Interventions and Measures:

* Ketamine low-dose infusion administered at 0.1 mg/kg/hr for 48 hours as an adjunct to standardized rib fracture management interventions as outlined in facility-approved Guidelines for Rib Fracture Management.
* The primary study outcome will be amount of narcotic used over the 48-hour study period (expressed as morphine mg equivalents).
* Secondary outcome measures will include: need for endotracheal intubation or non-invasive positive pressure ventilation, oxygen requirements, daily incentive spirometer values, daily forced vital capacity measurements, and subjective patient pain ratings.
* Other outcomes measured will be Intensive Care Unit stay, total hospital length of stay, and adverse medication effects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older
* Diagnosis of 3 or more acute rib fractures related to blunt traumatic chest injury.
* Able to undergo consent procedure and give valid consent, or availability of family member to provide consent for the study

Exclusion Criteria:

* Age <18 years
* Cognitively impaired
* Pregnant or lactating females.
* Glasgow Coma Score (GCS) of ≤ 14 at time of admission
* Evidence of increased intraocular pressure
* Presence of acute coronary syndrome
* Diagnosed moderate to severe traumatic brain injury
* Evidence of uncontrolled intracranial hypertension
* History of seizures or stroke
* History of severe psychiatric disorders
* Allergy to ketamine
* Currently being treated, prior to admission, with opiate agonist/antagonist therapy
* Presence of poorly controlled hypertension, cardiac arrhythmias, and/or tachycardia on admission
* Subjects who, in the opinion of the Investigator, may be inappropriate for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michaela A West, MD, PhD, Study Director — North Memorial Health; Joseph Farhat, MD, Principal Investigator — North Memorial Health
Locations (1):
- North Memorial Health Hospital, Robbinsdale, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walters MK, Farhat J, Bischoff J, Foss M, Evans C. Ketamine as an Analgesic Adjuvant in Adult Trauma Intensive Care Unit Patients With Rib Fracture. Ann Pharmacother. 2018 Sep;52(9):849-854. doi: 10.1177/1060028018768451. Epub 2018 Apr 2. PMID 29607659

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo/Control | Low Dose Ketamine Infusion (LDKI)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adult trauma in-patients with three or more rib fractures. Inclusion criteria were: age >18 years, known blunt chest trauma with >three rib fractures, and able to provide informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Control | Low Dose Ketamine Infusion (LDKI) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 17 | 30
  >=65 years | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (11.2) | 57.6 (14.8) | 62.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 17 | 20 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Average number fractured ribs [Mean (Standard Deviation); unit: Number of fractured ribs] | 5.7 (1.9) | 7.1 (3.8) | 6.3 (3.0)
Injury Severity Score (ISS) [Mean (Standard Deviation); unit: Units on a scale] — Injury Severity Score (ISS) is a summary descriptor of traumatic injuries derived from the three highest body region Abbreviated Injury Scores (AIS, range 1-6). The 3 highest AIS values are squared and added together to calculate ISS (ISS = A^2 + B^2 + C^2 where A, B, C are AIS scores of the 3 most injured ISS body regions). The ISS scores range from 1 to 75 (i.e. AIS scores of 5 for each category). Max score of 75 is considered "un-survivable". ISS value interpretation: 1-8 minor trauma, 9-15 moderate trauma, 16-24 severe trauma, greater than or equal to 25 very severe trauma.
  Units on a scale | 11.4 (3.2) | 15.1 (5.1) | 13.0 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Milligrams of Morphine Equivalents (MME) Administered
Description: Standardized method of reporting narcotic analgesic administration by converting opioid narcotics to the equivalent dosage of morphine that would yield same result.
Time Frame: Outcome was evaluated up to a total of 96 hours (from time zero to 48 hours of infusion and up to 48 hrs after infusion stopped.
Population: The Utah opioid morphine milligram equivalent conversion factor was used to convert all opioid analgesic doses administered during the study period.
Measure: Mean (Standard Deviation); unit: Morphine Milligam Equivalents (MME)
Arm/Group | Placebo/Control | Low Dose Ketamine Infusion (LDKI)
Number analyzed (Participants) | 25 | 25
Morphine Milligam Equivalents (MME) | 84.9 (31.9) | 81.7 (32.4)

2. Secondary Outcome: Pulmonary Complications
Description: Number of participants that develop pneumonia, require intubation, or non-invasive positive pressure ventilation
Time Frame: Up to 30 days after intervention (administration of study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Control | Low Dose Ketamine Infusion (LDKI)
Number analyzed (Participants) | 25 | 24
Participants
  Develop pneumonia | 3 | 0
  Require non-invasive positive pressure ventilation | 8 | 9
  Require intubation | 1 | 1
  No pulmonary complications | 13 | 14

3. Secondary Outcome: ICU Admission or Hospital Readmission
Description: Number of participants that requirie transfer to ICU (e.g., respiratory difficulty, tachycardia, hypotension, altered mental status) or that readmission to hospital after discharge for any reason.
Time Frame: Up to 30 days after intervention (administration of study drug)
Population: Unplanned intensive care unit (ICU) admission or hospital readmission for a condition related to rib fractures/chest trauma.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Control | Low Dose Ketamine Infusion (LDKI)
Number analyzed (Participants) | 25 | 24
Participants
  ICU Readmission within 30 days | 2 | 0
  Hospital Readmission within 30 days | 3 | 1
  No need for hospital or ICU readmission | 20 | 23

ADVERSE EVENTS:
Time Frame: Adverse events data were specifically analyzed for a time period within 30 days of initiation of study drug infusion.
Arm/Group | Placebo/Control | Low Dose Ketamine Infusion (LDKI)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/25
Other Adverse Events (participants affected / at risk) | 11/25 | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Control (N=25) | Low Dose Ketamine Infusion (LDKI) (N=25)
Acute Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Acute respiratory failure requring intubation and mechanical ventilation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Control (N=25) | Low Dose Ketamine Infusion (LDKI) (N=25)
Non-serious adverse events (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (9) — Development of pneumonia or non-life threatening lung complications up to 30 days after study drug infusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT06236113/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT06236113/ICF_002.pdf